CLINICAL TRIAL: NCT01970631
Title: The Study of Physical Activity Rewards After Knee Surgery
Acronym: SPARKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Elena Losina, Co-Director, Orthopaedic and Arthritis Center for Outcomes Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013P000916; R21AR063913 (NIH)
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis; Degenerative Joint Disease
Keywords: Osteoarthritis; Total Knee Replacement; total Knee Arthroplasty; Post-operative recovery TKR; Physical Activity; Motivational Interviewing; Financial Incentives
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Usual Care (No Intervention): Participants randomized to the Usual Care group will receive the current standard post-operative TKR care.
- Motivational Interviewing (MI) (Active Comparator): Participants randomized to the MI Intervention group will receive up to 14 telephone calls from a Health Educator for 9 months post-TKR.
  Interventions: Behavioral: Motivational Interviewing (MI)
- Financial Incentives (FI) (Active Comparator): Participants randomized to the FI Intervention group will receive financial incentives for completing physical activity logs weekly/bi-weekly and achieving pre-specified physical activity goals over the course of the study.
  Interventions: Other: Financial Incentives
- Motivational Inverterviewing (MI) + Financial Incentives (FI) (Active Comparator): Participants randomized to the FI + MI Intervention group will receive financial incentives for completing physical activity logs weekly/bi-weekly and achieving pre-specified physical activity goals as well as receive up to 14 telephone calls from a Health Educator for 9 months post-TKR.
  Interventions: Behavioral: Motivational Interviewing (MI); Other: Financial Incentives

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — The motivational interviewing arms of SPARKS will consist of Health Educators trained in Motivational Interviewing (MI) techniques contacting participants at regular intervals over the course of the nine months following participants' total knee replacement (TKR).
  Arms: Motivational Interviewing (MI); Motivational Inverterviewing (MI) + Financial Incentives (FI)
Other: Financial Incentives — The financial intervention arms of SPARKS will provide compensation to participants for completing physical activity logs weekly/bi-weekly and reaching pre-specified physical activity goals.
  Arms: Financial Incentives (FI); Motivational Inverterviewing (MI) + Financial Incentives (FI)

SUMMARY:
The objectives of this research are to conduct a proof of concept randomized controlled trial with 200 patients undergoing primary total knee replacement (TKR) at Brigham and Women's Hospital (BWH). The trial will compare levels of physical activity in subjects in the behavioral and economic interventions versus "Usual Care" post TKR.

DETAILED DESCRIPTION:
Physical activity (PA) has been shown to improve pain and function in persons with knee osteoarthritis (OA), reduce obesity, and prevent the onset and progression of heart disease, diabetes, and chronic pulmonary disease. The US Department of Human and Health Services (DHHS) guidelines recommend that adults engage in >150 minutes of moderate physical activity per week. However, adherence to PA guidelines is poor in the general population, particularly in persons with knee OA.

Total knee replacement (TKR) is widely used in patients with symptomatic, advanced knee OA. While the vast majority of persons undergoing TKR experience considerable reduction in pain and improvement in functional capacity, far fewer take this opportunity to become more physically active. Since physical activity has a direct relationship with quality of life and with prevention and amelioration of many chronic conditions, many TKR recipients do not derive maximum benefits from the procedure.

The focus of this proposal is to conduct a proof of concept RCT to establish the efficacy of a behavioral economics-based intervention that would facilitate engagement in physical activity and improve adherence to PA guidelines in the growing population of TKR recipients. We address the innovative hypothesis that the period following TKR presents a window of opportunity to fundamentally change attitudes and beliefs regarding PA, and that tangible economic incentives will effectively induce behavior change and facilitate adherence to PA guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary TKA at BWH
* Osteoarthritis is the principal underlying diagnosis
* Age >=40 at the projected date of TKA
* English-speaking
* Willing and able to access the internet to complete study related questionnaires

Exclusion Criteria:

* Osteoarthritis is not the principal underlying diagnosis (e.g. inflammatory arthritis)
* Dementia (can not fill out forms)
* Psychological issues that preclude participation, as identified by participating surgeons
* Does not have access to a computer and/or the internet.
* Non-English speaker (instruments are not validated in Spanish); very few non-English speakers (<5%) are otherwise eligible
* Age <40 at the projected date of TKA (TKA is usually due to major trauma, juvenile onset or congenital disease)
* Lives in a nursing home (difficult to track costs)
* Implantation of Unicompartamental Knee Arthroscopy (different clinical features and different costs)
* Bilateral TKA in same admission (simultaneous), staged or within 6 months
* Uses a wheelchair or walker to ambulate
* Has been told by a physician that he/she has a heart condition and should only do physical activity recommended by a doctor
* Has pain in his/her chest when doing physical activity
* Loses balance because of dizziness
* Loses consciousness
* Unable/unwilling to wear Fitbit® accelerometer for 5 or more days during baseline visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-01-09 (Actual); Primary Completion 2016-11-05 (Actual); Study Completion 2016-11-05 (Actual)

PRIMARY OUTCOMES:
number of steps | 6 months
  The primary outcome is the average number of steps over 7 days as measured by accelerometer at 6 months post-TKR.

SECONDARY OUTCOMES:
Adherence to PA guidelines | 6-months
  The secondary outcome will be adherence to PA guidelines, defined by the DHHS as >150 minutes of moderate or greater intensity PA occurring in bouts of 10 minutes or more per week.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Losina, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Losina E, Collins JE, Deshpande BR, Smith SR, Michl GL, Usiskin IM, Klara KM, Winter AR, Yang HY, Selzer F, Katz JN. Financial Incentives and Health Coaching to Improve Physical Activity Following Total Knee Replacement: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 May;70(5):732-740. doi: 10.1002/acr.23324. Epub 2018 Apr 12. PMID 28732147
- [Derived] Usiskin IM, Yang HY, Deshpande BR, Collins JE, Michl GL, Smith SR, Klara KM, Selzer F, Katz JN, Losina E. Association between activity limitations and pain in patients scheduled for total knee arthroplasty. BMC Musculoskelet Disord. 2016 Sep 1;17(1):378. doi: 10.1186/s12891-016-1233-2. PMID 27585441